CLINICAL TRIAL: NCT01547039
Title: Platelet Reactivity Testing in Association With Perioperative Microembolic Signals During Carotid Endarterectomy
Brief Title: Platelet Reactivity and MES During CEA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Gert Jan de Borst, MD, PhD, UMC Utrecht
Other Study IDs: NL33061.051.10
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Carotid Artery Stenosis; Ischemic Stroke; Myocardial Infarction; Aspirin Resistance
Keywords: Carotid endarterectomy; Transcranial doppler; Micro embolic signals; Platelets; Aspirin
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid endarterectomy (CEA): Patients undergoing carotid endarterectomy

SUMMARY:
The purpose of this study is to analyze the association between aspirin efficacy and general platelet reactivity in relation to microembolic signals (MES) during carotid endarterectomy (CEA).

ELIGIBILITY:
Inclusion Criteria:

* Al patients undergoing elective carotid endarterectomy

Exclusion Criteria:

* Patients requiring a blood transfusion prior to surgery
* Patients with an inappropriate temporal bone window for transcranial Doppler (TCD)
* Patients on vitamin K antagonists or antiplatelet treatment other then aspirin
* Patients with an artificial cardiac valve

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective carotid endarterectomy in University Medical Centre Utrecht
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Microembolic signals (MES) | During and 1 hour following carotid endarterectomy (CEA)
  Microembolic signals detected by transcranial duplex (TCD)

SECONDARY OUTCOMES:
Ischemic stroke | within 30 days postoperative
Asymptomatic perioperative myocardial injury | 3 days postoperative
  Troponin elevation > 0.1 ng/ml
Myocardial infarction | Within 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gert Jan de Borst, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands